CLINICAL TRIAL: NCT01403467
Title: Impact of Continuous Positive Airway Pressure on the Treatment of Acute Asthma Exacerbation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Dr.Yuda Sutherasan, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-52-28; MURA2009/1239 (Other: Ramathibodi Hospital)
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2010-12

CONDITIONS: Acute Asthma
Keywords: Bronchial disease; asthma; continuous positive airway pressure (CPAP); Bronchoconstriction
MeSH Terms: conditions — Bronchial Diseases; Asthma | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NIPPV (Experimental)
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Device: Continuous positive airway pressure — CPAP 8 cmH2O
  Other Names: GoodKnight 420 G; Nellcor Puritan Bennett Inc.

SUMMARY:
This current study aimed to demonstrate the effectiveness of the addition of CPAP to the current conventional therapy in terms of airway obstruction improvement in acute asthma patients.

DETAILED DESCRIPTION:
Continuous positive airway pressure (CPAP) is widely used in providing ventilator support. However, its role in an acute asthmatic attack is uncertain. The purpose of this study was to compare the efficacy of CPAP when used in addition to conventional therapy with conventional therapy alone in the management of acute asthma exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years
* known asthmatic patients visiting ED with acute exacerbation
* had given their written informed consent.

Exclusion Criteria:

* smoking history
* chronic obstructive pulmonary disease
* required intubation
* instability of hemodynamic or arrhythmia
* unable to perform PEFR
* facial abnormality
* pulmonary infiltration
* pregnancy.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
an improvement in PEFR, as % predicted | 75 mins

CONTACTS AND LOCATIONS:
Overall Officials: Yuda Sutherasan, M.D., Principal Investigator — Ramathibodi Hospital, Mahidol University
Locations (1):
- Ramathibodi Hospital, Bangkok, Thailand